CLINICAL TRIAL: NCT03203356
Title: Evaluation of Adrenal Function Before and After GH Treatment in GHD Affected by GH Deficiency
Brief Title: Adrenal Function in GHD Children
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Carla Giordano, Prof. Carla Giordano, University of Palermo
Other Study IDs: UPalermo ITT-GHD
Record Dates: First submitted 2017-05-26; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Growth Hormone Treatment; Adrenal; Functional Disturbance
Keywords: growth hormone; children; adrenal function
MeSH Terms: interventions — Growth Hormone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GHD children: about 30 prepubertal children affected by overt idiopathic GHD
  Interventions: Drug: growth hormone
- controls: about 30 prepubertal children with constitutional short stature without endocrine disease

INTERVENTIONS:
Drug: growth hormone — Children with a diagnosis of GHD will practice GH replacement therapy in line with normal clinical practice and international guidelines. Controls will be evaluated just at baseline.
  Groups: GHD children

SUMMARY:
To evaluate in children affected by idiopathic GHD the adrenal function both at baseline and after 6 and 12 months of GH treatment.

DETAILED DESCRIPTION:
The relationship between the growth hormone (GH)-insulin like growth factor (IGF)-I system and the hypothalamic-pituitary-adrenal (HPA) axis is complex and not univocal. Both a stimulatory and neutral effect of IGF-I on HPA axis has been demonstrated in in vitro models and in healthy subjects, respectively. The effect of GH on the 11beta-hydroxysteroid dehydrogenases (11beta-HSD) isozymes is always to be considered in patients affected by GHD both at diagnosis and during GH treatment. Indeed, in peripheral tissues, corticosteroid hormone action is partially determined by the activity of 11beta-HSD, two isozymes of which interconvert hormonally active cortisol and inactive cortisone. 11beta-HSD2 inactivates cortisol to cortisone in the kidney, whilst 11beta-HSD1 performs the reverse reaction activating cortisol from cortisone in the liver and adipose tissue.

For these reasons, many data are available about the evaluation of adrenal function in patients affeceted byGHD, but most of them come from patients with organic GHD or adult patients, while few and discordant data are available on pediatric GHD patients. We aimed to evaluate, through insulin tolerance test, the adrenal function in about 30 children with overt diagnosis of idiopathic GHD both at baseline and after 6 and 12 months of GH treatment.

ELIGIBILITY:
Inclusion Criteria:

* prepubertal children with overt idiopathic growth hormone deficiency

Exclusion Criteria:

* Children with organic growth hormone deficiency or under treatment with glucocorticoids

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 30 consecutive children with short stature and overt idiopathic GHD and 30 children with constitutional short stature without endocrine disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of adrenal function in GHD children at baseline and in control group | baseline
  We will evaluate through insulin tolerance test the response of serum cortisol levels in GHD children at diagnosis (before start of GH therapy) and in controls subjects
Change in adrenal function in GHD children during GH therapy | 6 and 12 months
  We will evaluate through insulin tolerance test the response of serum cortisol levels in GHD children after 6 and 12 months of GH therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Endocrinology - University of Palermo, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No
IPD will be available just for our study